CLINICAL TRIAL: NCT00983905
Title: A One-Directional, Open-Label, Drug Interaction Study to Investigate the Effects of Multiple-Dose Colchicine on Single-Dose Pharmacokinetics of Theophylline in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study of Colchicine and Theophylline
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1010
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Pharmacokinetics
Keywords: healthy;; adult;; blood levels over time
MeSH Terms: interventions — Theophylline; Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Theophylline alone (Active Comparator): baseline theophylline kinetics
  Interventions: Drug: Theophylline
- Theophylline with steady-state Colchicine (Experimental): theophylline pharmacokinetics upon administration with colchicine at steady-state
  Interventions: Drug: Theophylline; Drug: Colchicine

INTERVENTIONS:
Drug: Theophylline — single doses of 300 mg (80 mg/15 ml elixer) administered alone at 7:45 am on Day 1 and then along with colchicine at 7:45 am on Day 19
  Other Names: Elixophyllin® Elixir (Theophylline Anhydrous) 80/15 ml concentrate
Drug: Colchicine — one 0.6 mg tablet twice daily at 7:45 am and 7:45 pm on Days 5 to 19
  Arms: Theophylline with steady-state Colchicine

SUMMARY:
Colchicine is a supressor of hepatic CYP1A2 and theophylline is a sensitive CYP1A2 probe substrate. When the two are co-administered the potential exists for a clinically significant drug interaction. This study aims to determine the effect of steady-state colchicine on the pharmacokinetics of theophylline administered as a single dose. A secondary goal is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the entire study period.

DETAILED DESCRIPTION:
Colchicine is a supressor of hepatic CYP1A2 and theophylline is a sensitive CYP1A2 probe substrate. When the two are co-administered the potential exists for a clinically significant drug interaction . This study aims to determine the effect of steady-state colchicine on the pharmacokinetics of theophylline administered as a single dose. After a fast of at least 10 hours, thirty healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one dose of 300mg (80mg/15ml concentrate) theophylline (theophylline elixir) on Day 1. Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately determine the pharmacokinetics of theophylline. Blood sampling will then continue on a non-confined basis on days 2-3. A four day washout period will be completed after the theophylline dose on Day 1 and prior to administration of the first colchicine dose on Day 5. Participants will return to the clinic on days 5-18 for non-confined dosing of colchicine (0.6mg every 12 hours). Administered dosing on these days will not necessarily be in a fasted state.

On Day 19 after a fast of at least 10 hours, all study participants will receive 300mg theophylline (80mg/15ml) and 0.6 mg colchicine (1 x 0.6mg tablet) together. Fasting will continue for 4 hours following these co-administered doses. All subjects will be confined to the clinic for dosing and the following 24-hour period. Blood samples will be drawn at times sufficient to adequately determine the pharmacokinetics of theophylline in the presence of colchicine at steady state. Blood sampling will continue on a non-confined basis on Days 20-21. The final dose of colchicine (1x0.6mg) will be administered to subjects the evening of Day 19.

A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse will be measured prior to dosing and at approximately 1, 2, and 3 hours following drug administration on Days 1, 5 (after the morning dose) and 19. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (postmenopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or donation of plasma
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-08; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty (30) healthy, non-smoking, male and female volunteers, consisting of members of the community at large, were to be enrolled.
Pre-assignment Details: 44 subjects screened, 6 were screen failures, 8 had schedule conflicts
Groups:
- Theophylline Alone / With Colchicine (at Steady State): [All subjects received each of the study treatments.] Each subject received a single 300 mg dose of theophylline elixer (80 mg/15 ml concentrate) on Day 1 at 7:45am after an overnight fast of at least 10 hours, followed by a washout period of 4 days. On Days 5 to 18, each subject received one 0.6 mg colchicine tablet twice daily at 7:45am and 7:45pm without regard to meals. Then, on Day 19, each subject received both a single dose of theophylline elixer (80 mg/15 ml concentrate) and one 0.6 mg colchicine tablet at 7:45am after an overnight fast of at least 10 hours. (They also received the final dose of one 0.6 mg colchicine tablet at 7:45 pm.)
Period: Theophylline Alone
Arm/Group | Theophylline Alone / With Colchicine (at Steady State)
Started | 30
Completed | 29 (withdrawn by sponsor due to vomiting(1))
Not Completed | 1
Not completed — Adverse Event | 1
Period: 4 Day Washout Period
Arm/Group | Theophylline Alone / With Colchicine (at Steady State)
Started | 29
Completed | 29
Not Completed | 0
Period: Colchicine Alone
Arm/Group | Theophylline Alone / With Colchicine (at Steady State)
Started | 29
Completed | 27 (withdrawn by sponsor due to: diarrhea(1); vomiting and diarrhea(1))
Not Completed | 2
Not completed — Adverse Event | 2
Period: Theophylline With Colchicine
Arm/Group | Theophylline Alone / With Colchicine (at Steady State)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Theophylline Alone / With Colchicine (at Steady State)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants] — age range: >=18 and <=45 years old
  Participants
    <=18 years | 2
    Between 18 and 65 years | 28
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 25.1 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that theophylline drug reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn within 1 hour prior to theophylline dosing (0 hour) on Days 1 and 19, then at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36, and 48 hours after theophylline dose administration
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Theophylline Alone: On Day 1, each subject received a single 300 mg dose of theophylline elixer (80 mg/15 ml concentrate) at 7:45 am after an overnight fast of at least 10 hours, followed by a washout period of 4 days.
- Theophylline With Colchicine (at Steady-state): On Days 5 to 18, each subject received one 0.6 mg colchicine tablet twice daily at 7:45 am and 7:45 pm without regard to meals. Then, on Day 19, each subject received both a single dose of theophylline elixer (80 mg/15 ml concentrate) and one 0.6 mg colchicine tablet at 7:45am after an overnight fast of at least 10 hours. (They also received the final dose of one 0.6 mg colchicine tablet at 7:45 pm.)
Arm/Group | Theophylline Alone | Theophylline With Colchicine (at Steady-state)
Number analyzed (Participants) | 27 | 27
µg/mL | 9.76 (2.25) | 9.79 (1.87)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the theophylline plasma concentration versus time curve, from time 0 to the time of the last measurable theophylline concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg-hr/mL
Arm/Group | Theophylline Alone | Theophylline With Colchicine (at Steady-state)
Number analyzed (Participants) | 27 | 27
µg-hr/mL | 120.80 (38.73) | 121.35 (40.06)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the theophylline plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable theophylline plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg-hr/mL
Arm/Group | Theophylline Alone | Theophylline With Colchicine (at Steady-state)
Number analyzed (Participants) | 27 | 27
µg-hr/mL | 127.47 (42.28) | 129.39 (44.83)

ADVERSE EVENTS:
Groups:
- Theophylline Alone: Each subject received a single 300 mg dose of theophylline elixer (80 mg/15 ml concentrate) on Day 1 at 7:45 am after an overnight fast of at least 10 hours, followed by a washout period of 4 days.
- Colchicine Alone: On Days 5 to 18, each subject received one 0.6 mg colchicine tablet twice daily at 7:45 am and 7:45 pm without regard to meals.
- Theophylline With Steady-state Colchicine: On Day 19, each subject received both a single dose of theophylline elixer (80 mg/15 ml concentrate) and one 0.6 mg colchicine tablet at 7:45 am after an overnight fast of at least 10 hours. (They also received the final dose of one 0.6 mg colchicine tablet at 7:45 pm.)
Arm/Group | Theophylline Alone | Colchicine Alone | Theophylline With Steady-state Colchicine
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 8 | 15 | 6
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Theophylline Alone | Colchicine Alone | Theophylline With Steady-state Colchicine
ear discomfort (Ear and labyrinth disorders) | 0/30 (0) | 1/29 (1) | 0/27 (0)
eye pruritus (Eye disorders) | 1/30 (1) | 0/29 (0) | 0/27 (0)
abdominal pain (Gastrointestinal disorders) | 1/30 (1) | 1/29 (2) | 1/27 (1)
abdominal pain upper (Gastrointestinal disorders) | 0/30 (0) | 3/29 (3) | 0/27 (0)
diarrhoea (Gastrointestinal disorders) | 0/30 (0) | 8/29 (11) | 0/27 (0)
dyspepsia (Gastrointestinal disorders) | 0/30 (0) | 1/29 (1) | 0/27 (0)
nausea (Gastrointestinal disorders) | 5/30 (7) | 2/29 (3) | 0/27 (0)
stomach discomfort (Gastrointestinal disorders) | 0/30 (0) | 1/29 (1) | 0/27 (0)
vomiting (Gastrointestinal disorders) | 1/30 (1) | 3/29 (3) | 1/27 (2)
feeling hot (General disorders) | 0/30 (0) | 1/29 (2) | 0/27 (0)
skin laceration (Injury, poisoning and procedural complications) | 0/30 (0) | 1/29 (1) | 0/27 (0)
heart rate increased (Investigations) | 0/30 (0) | 0/29 (0) | 1/27 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 0/30 (0) | 0/29 (0) | 1/27 (1)
dizziness (Nervous system disorders) | 3/30 (4) | 4/29 (5) | 2/27 (2)
headache (Nervous system disorders) | 2/30 (2) | 3/29 (4) | 2/27 (2)
paraesthesia (Nervous system disorders) | 0/30 (0) | 0/29 (0) | 1/27 (1)
syncope (Nervous system disorders) | 0/30 (0) | 0/29 (0) | 1/27 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/30 (1) | 0/29 (0) | 0/27 (0)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/30 (0) | 1/29 (1) | 0/27 (0)
drug eruption (Skin and subcutaneous tissue disorders) | 1/30 (1) | 0/29 (0) | 0/27 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days